CLINICAL TRIAL: NCT02047188
Title: Observation of Microvessels and Invasion in Early Colorectal Lesions by Narrow Band Imaging:Combination With Microvessel Count and MMP-7 Expression
Brief Title: Observation of Microvessels and Invasion in Early Colorectal Lesions by NBI
Status: Completed | Type: Observational
Sponsor: Xiaobo Li (Other)
Responsible Party: Sponsor-Investigator, Xiaobo Li, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Organization: Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: 12YZ036
Record Dates: First submitted 2014-01-25; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Colorectal Neoplasms
Keywords: narrow band imaging,microvessels,matrix metalloproteinase-7
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Samples after biopsy or resection are to be retained.
Oversight: Data Monitoring Committee: No

SUMMARY:
Combined with magnifying endoscopy,narrow-band imaging (NBI) contrasts microvascular architecture on lesion surface.The histology of early colorectal lesions could be predicted under NBI view.However,its capability for estimating invasion depth remains to be verified.The study is based on the hypothesis:NBI can predict histology and invasion depth,combined with the verification of microvessel count and MMP-7 expression.

DETAILED DESCRIPTION:
The microvessel count (MVC) is a classical method of assessing histologic grade.To verify whether NBI could predict histology through microvascular architecture,we measured lesion microvessels by immunohistochemistry.On the other hand,we applied immunohistochemistry of matrix metalloproteinase-7 (MMP-7) to validate the capability of NBI for estimating invasion depth.MMP-7 is directly involved in the processes of growth, invasion, and metastasis of colorectal cancer.Our target was to clarify the diagnostic accuracy of magnifying NBI in early colorectal lesions,combined with the verification of microvessel count and MMP-7 expression.

ELIGIBILITY:
Inclusion Criteria:

* patients of early colorectal lesions with capillary pattern(CP) type II&III,initially detected by white-light view and then examined by NBI with magnifying endoscopy.

Exclusion Criteria:

* lesions with CP type I;
* CP type III lesions with an obvious appearance of advanced cancer;
* lesions that had underwent biopsy;
* patients with inflammatory bowel disease(IBD) or familial adenomatous polyposis(FAP)
* patients with previous colorectal surgery;
* having conditions associated with cardiac,hepatic,renal,and coagulopathy diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with early colorectal lesions
Sampling Method: Non-Probability Sample
Enrollment: 418 (Actual)
Dates: Start 2010-01; Primary Completion 2013-05 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
NBI prediction for lesion histology and invasion | in two weeks after lesion treatment
  We will receive the histologic findings in two weeks after lesion treatment.Then we can compare NBI prediction with the final histologic type.

SECONDARY OUTCOMES:
immunohistochemical outcome of microvessel count and MMP-7 | in three days after immunohistochemistry
  We will receive the immunohistochemical outcome in three days after immunohistochemistry.Then we can compare NBI prediction with immunohistochemical outcome

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobo Li, Ph.D, Principal Investigator — Shanghai Ren Ji Hospital